CLINICAL TRIAL: NCT04320849
Title: Human Use Condition Study-Fluoroscopic Evaluation of 3D Curvature of Implanted Right Ventricular Leads in Humans
Brief Title: Human Use Condition Study- Evaluation of Implanted Leads in Humans
Acronym: HUCS
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Abbott (Industry); Medtronic (Industry); Biotronik SE & Co. KG (Industry); Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00103284
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Results first posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Pacemaker Malfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with protocol identified RV Leads: Medtronic model 6935M (Quattro Secure Single Coil Defibrillation Lead) Abbott model LDA 210Q (Optisure Single Coil Defibrillation Lead) Abbott model LDA 220Q (Optisure Dual Coil Defibrillation Lead) Boston Scientific model 4470/4471 (FINELINE II/FINELINE II Sterox); Positive Fixation Biotronik model Solia S (Active Fixation Leads)

SUMMARY:
The purpose of this study is to evaluate different types of leads (wires) that are connected to your pacemaker (an implanted device which assists your heart function) to understand how the shape and motion of your previously implanted lead changes in the body.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate different types of leads (wires) that are connected to the pacemaker (an implanted device which assists enrolled subject's heart function) to understand how the shape and motion of the previously implanted lead changes in the body.

ELIGIBILITY:
Inclusion Criteria:

Patients with RV leads included in the scope of this study whose system has been implanted for at least 3 calendar months Patients at least 18 years of age and capable of providing informed consent Patients who can physically perform range of arm motion and breath-holding described in the imaging protocol Patients who are willing and able to comply with instruction related to the imaging protocol

Exclusion Criteria:

Planned lead modification Patients with abandoned leads (includes: RV/RA/LV) Patients undergoing second or subsequent pulse generator change Patient has permanent atrial arrhythmias Limited life expectancy or medical condition that would not allow completion of the study Patient is known to be pregnant or breastfeeding at time of consent Limited range of mobility of the implant location arm Patient is unable to climb on and off an examination table unassisted Patients deemed hemodynamically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll at least 80 and up to 120 subjects with one of four different specified market-released lead families. The leads are from all four CIED manufacturers participating in this protocol. Approximately 30 leads from each manufacturer's lead family will be required.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Piccini, MD, Principal Investigator — Duke University
Locations (5):
- United States (5):
  - Cedars Sinai Medical Center, Los Angeles, California
  - MercyOne Iowa Heart Center, Des Moines, Iowa
  - Minneapolis Heart Institute, Saint Paul, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - Trinity Clinic, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Consented Patients With RV Pacing Leads and Defibrillation Leads: Defibrillation leads consisted of the following:
  Manufacturer: Abbott Model: LDA 210Q Description: Optisure Single Coil Defibrillation Lead
  Manufacturer: Abbott Model: LDA 220Q Description: Optisure DualCoil Defibrillation Lead Number of Leads Imaged: 8
  Manufacturer: Medtronic Model: 6935M Description: Quattro Secure Single Coil Defibrillation Lead
  Manufacturer: Biotronik Model: Solia S Description: Active Fixation Leads
  Manufacturer: Boston Scientific Model: 4470 Description: FINELINE II/FINELINE II Sterox EZ Positive Fixation (polyurethane)
  Manufacturer: Boston Scientific Model: 4471 Description: FINELINE II/FINELINE II Sterox EZ Positive Fixation (polyurethane)
Period: Overall Study
Arm/Group | Consented Patients With RV Pacing Leads and Defibrillation Leads
Started | 117
Completed | 109
Not Completed | 8
Not completed — Withdrawal by Subject | 4
Not completed — Imaging data unavailable | 2
Not completed — Incomplete imaging | 2

BASELINE CHARACTERISTICS:
Groups:
- Consented Patients With RV Pacing Leads and Defibrillation Leads: Defibrillation leads consisted of the following:
  Manufacturer: Abbott Model: LDA 210Q Description: Optisure Single Coil Defibrillation Lead Number of Leads Imaged: 21
  Manufacturer: Abbott Model: LDA 220Q Description: Optisure DualCoil Defibrillation Lead Number of Leads Imaged: 8
  Manufacturer: Medtronic Model: 6935M Description: Quattro Secure Single Coil Defibrillation Lead Number of Leads Imaged: 27
  Manufacturer: Biotronik Model: Solia S Description: Active Fixation Leads Number of Leads Imaged: 23
  Manufacturer: Boston Scientific Model: 4470 Description: FINELINE II/FINELINE II Sterox EZ Positive Fixation (polyurethane) Number of Leads Imaged: 1
  Manufacturer: Boston Scientific Model: 4471 Description: FINELINE II/FINELINE II Sterox EZ Positive Fixation (polyurethane) Number of Leads Imaged: 31
Arm/Group | Consented Patients With RV Pacing Leads and Defibrillation Leads
Number analyzed (Participants) | 117
Age, Continuous [Mean (Full Range); unit: years] | 68.72 [30.58 to 93.28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 105
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 17
  White | 94
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 117

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With in Vivo Cyclic Mean Curvature of Pacing and Defibrillation Leads in the Extravenous Region Determined During Specified Arm Movements
Description: Measure dynamic in vivo curvature of RV pacing and defibrillator leads in the extravenous and intracardiac anatomy
  ***In vivo cyclic mean curvature of RV pacing and defibrillation leads in the extravenous region will be determined during specified arm movements. The relationship between lead stiffness and curvature will be evaluated.
Time Frame: Approximately 1 month
Population: Consented patients with imaging data.
Measure: Count of Participants; unit: Participants
Arm/Group | Consented Patients With RV Pacing Leads and Defibrillation Leads
Number analyzed (Participants) | 109
Participants | 109
Statistical Analysis 1: Comparison: Consented Patients With RV Pacing Leads and Defibrillation Leads; The following set of hypotheses were used to evaluate the relationship between lead stiffness and curvature in the extravenous region: H0: a ≥ 0 Ha: a < 0 where a represents the coefficient for stiffness in the following model: log (curvature) = a*stiffness + b + normally distributed error; Test type: Other; Slope = 0.0675, 90% CI 1-sided [upper limit 0.106]

2. Primary Outcome: Number of Participants With in Vivo Cyclic Mean Curvature of Pacing and Defibrillation Leads in the Intracardiac Region Determined During Two or More Cardiac Cycles
Description: Measure the relationship between lead bending stiffness and in vivo curvature
  ***In vivo cyclic mean curvature of RV pacing and defibrillation leads in the intracardiac region will be determined during two or more cardiac cycles. The relationship between lead stiffness and curvature will be evaluated.
Time Frame: Approximately 1 month
Population: Consented patients with imaging data.
Measure: Count of Participants; unit: Participants
Arm/Group | Consented Patients With RV Pacing Leads and Defibrillation Leads
Number analyzed (Participants) | 109
Participants | 109
Statistical Analysis 1: Comparison: Consented Patients With RV Pacing Leads and Defibrillation Leads; The following set of hypotheses will be used to evaluate the relationship between lead stiffness and curvature in the intracardiac region: H0: a ≥ 0 Ha: a < 0 where a represents the coefficient for stiffness in the following model: log (curvature) = a*stiffness + b + normally distributed error; Test type: Other; Slope = 0.199, 90% CI 1-sided [upper limit 0.397]

3. Primary Outcome: Number of Participants With in Vivo Cyclic Mean Curvature of Pacing and Defibrillation Leads in the Connector Region Determined During Specified Arm Movements
Description: Assess the relationship between subject and implant variables and lead curvature
  ***In vivo cyclic mean curvature of RV pacing and defibrillation leads in the connector region were determined during specified arm movements. The relationship between lead stiffness and curvature was evaluated.
Time Frame: Approximately 1 month
Population: Consented patients with imaging data.
Measure: Count of Participants; unit: Participants
Arm/Group | Consented Patients With RV Pacing Leads and Defibrillation Leads
Number analyzed (Participants) | 109
Participants | 109
Statistical Analysis 1: Comparison: Consented Patients With RV Pacing Leads and Defibrillation Leads; The following set of hypotheses were used to evaluate the relationship between lead stiffness and curvature in the connector region: H0: a ≥ 0 Ha: a < 0 where a represents the coefficient for stiffness in the following model: log (curvature) = a*stiffness + b + normally distributed error; Test type: Other; Slope = -0.015, 90% CI 1-sided [upper limit 0.0123]

ADVERSE EVENTS:
Time Frame: 30 days from imaging
Groups:
- Consented Patients With RV Pacing Leads and Defibrillation Leads: Medtronic model 6935M (Quattro Secure Single Coil Defibrillation Lead) Abbott model LDA 210Q (Optisure Single Coil Defibrillation Lead) Abbott model LDA 220Q (Optisure Dual Coil Defibrillation Lead) Boston Scientific model 4470/4471 (FINELINE II/FINELINE II Sterox); Positive Fixation Biotronik model Solia S (Active Fixation Leads)
Arm/Group | Consented Patients With RV Pacing Leads and Defibrillation Leads
All-Cause Mortality (participants affected / at risk) | 0/117
Serious Adverse Events (participants affected / at risk) | 0/117
Other Adverse Events (participants affected / at risk) | 0/117

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT04320849/Prot_SAP_000.pdf